CLINICAL TRIAL: NCT02296372
Title: Pilot Observation of Continuous Glucose Monitoring in Critically Ill Patients Under Consideration of Accuracy, Feasibility and Acceptance by Ward Staff
Brief Title: Accuracy, Feasibility and Acceptance of Continuous Glucose Monitoring in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Steffen Weber-Carstens, PD Dr. med. Steffen Weber-Carstens, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Charité-MOTAFEE-CGM
Record Dates: First submitted 2014-11-04; First posted 2014-11-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Glucose Metabolism Disorders; Diabetic Blood Glucose Monitoring; Critical Illness
MeSH Terms: conditions — Glucose Metabolism Disorders; Critical Illness | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOFA <7 (Other): Critically ill patients with a Sequential Organ Failure Assessment (SOFA) score < 7 at first day of measurement.
  Intervention: Measuring continuous glucose monitoring.
  Interventions: Device: Continuous glucose monitoring
- SOFA >7 (Other): Critically ill patients with a Sequential Organ Failure Assessment (SOFA) score > 7 at first day of measurement.
  Intervention: Measuring continuous glucose monitoring.
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring by subcutaneous or intravasal device for 72 hours.
  In use MEDTRONIC SENTRINO® and Edwards GlucoClear® systems.
  Other Names: CGM

SUMMARY:
Critically ill patients are on high risk for increased serum glucose levels, leading to more comorbidity and higher mortality risk. In patients with severe sepsis and septic shock hyperglycemia is a typical finding. However the need of insulin therapy is associated with an increased risk of hypoglycemia. Newly developed technologies for continuous glucose monitoring in critically ill patients may improve glycemic control and reduce glucose variability. The investigators will perform continuous glucose monitoring in critically ill patients on ICU. Measurements will be done for a period of 72h per patient. The investigators aim is to evaluate accuracy feasibility and acceptance of these methods. To analyze accuracy sensor glucose levels will be validated due to arterial blood gas measurements with the blood gas analyzer. The investigators will investigate the influence of several factors like oedema, perspiration, BMI, body temperature, pH-value application of vasoconstrictors on accuracy and feasibility of the particular system. Furthermore Nursing staff will be given a questionnaire to identify acceptance.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients with expected ICU stay for more than 72 hours
* informed consent by the patients or legal proxy

Exclusion Criteria:

* age < 18
* no informed consent by the patients or legal proxy
* pregnancy
* infaust prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of continuous glucose monitoring compared to blood gas analyses | 72 hours
  Difference between glucose values of continuous glucose monitoring and blood gas analyses

SECONDARY OUTCOMES:
Feasibility of continuous glucose monitoring | 72 hours
  Problems within the application of sensor and monitoring during ward routine
Acceptance of continuous glucose monitoring by physicians and nursing staff | 72 hours
  Acceptance and evaluation of the device by physicians and nursing staff evaluated by questionnaire

OTHER OUTCOMES:
Technical problems with the monitoring | up to 72 hours
  Number of needed sensors per patient. Duration of functional sensor. Number and reasons for accidentally sensor removal.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Weber-Carstens, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

REFERENCES:
- [Result] Wollersheim T, Engelhardt LJ, Pachulla J, Moergeli R, Koch S, Spies C, Hiesmayr M, Weber-Carstens S. Accuracy, reliability, feasibility and nurse acceptance of a subcutaneous continuous glucose management system in critically ill patients: a prospective clinical trial. Ann Intensive Care. 2016 Dec;6(1):70. doi: 10.1186/s13613-016-0167-z. Epub 2016 Jul 21. PMID 27439710